CLINICAL TRIAL: NCT01319682
Title: Intravenous Lidocaine for Effective Pain Relief After Posterior Lumbar Spinal Fusion: a Prospective, Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Effect of Intravenous Lidocaine on Pain After Lumbar Spinal Fusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Hyun Kang, Assistant professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChungAngUH2
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Pain
Keywords: Pain; Preemptive; Lidocaine; Intravenous; Lumbar fusion
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous lidocaine injection group (Active Comparator): Patients in Group I (intravenous lidocaine injection group) received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.
  Interventions: Drug: Intravenous lidocaine injection
- Placebo control group (Placebo Comparator): Patients in Group C (placebo control group) received normal saline intravenous injection
  Interventions: Drug: Intravenous normal saline injection

INTERVENTIONS:
Drug: Intravenous lidocaine injection — Patients in Group I (intravenous lidocaine injection group) received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.
  Other Names: IV lidocaine
  Arms: Intravenous lidocaine injection group
Drug: Intravenous normal saline injection — The patients in Group C (placebo control group) received normal saline intravenous injection
  Other Names: IV saline
  Arms: Placebo control group

SUMMARY:
This prospective randomized study aims to evaluate the effectiveness of intravenous lidocaine injection on the relief of pain in patients undergoing 1-level posterior lumbar fusion.

A total of 54 patients will be randomized into one of two groups (group C or group I) based on Excel number generation.

Patients in group C will receive received normal saline intravenous injection, and patients in group I will receive an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.

Visual analogue scale pain scores, fentanyl consumption and the frequency at which patients pushed the button (FPB) of a patient-controlled analgesia system will be recorded at 4, 12, 24, 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 1-level posterior lumbar fusion

Exclusion Criteria:

* mental change
* allergy to local anesthetics
* chronic analgesics user

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Postopeartive pain measured using Visual analogue scale at postoperative 4hour | post op 4hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 4hour.

SECONDARY OUTCOMES:
visual analogue scale 12 hour | Post op 12 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 12 hour.
visual analogue scale 24hour | Post op 24 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 24 hour.
Visual analogue scale 48hour | Post Op 48hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 48 hour.
Opioid consumption 4hour | Post Op 4hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 4hour will be measured.
Opioid consumption 24hour | Post op 24 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid from 12 hour to post op 24 hour will be measured.
Opioid consumption 12 hour | Post Op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid from post op 4hour to post op 12 hour will be measured.
Opioid consumption 48hour | Post Op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid from post op 24 hour to post op 48 hour will be measured
FPB 4 hour | Post Op 4 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 4 hour will be measured.
FPB 12 hour | post op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) from post op 4 hour to post op 12 hour will be measured.
FPB 24 hour | Post Op 24 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) fom post op 12 hour to post op 24 hour will be measured.
FPB 48 hour | Post Op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) fom post op 24 hour to post op 48 hour will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kang, Ph.D.,, Study Chair — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Young-Baeg Kim, Ph.D., Study Director — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- ChungAng University, Seoul, South Korea

REFERENCES:
- [Derived] Kim KT, Cho DC, Sung JK, Kim YB, Kang H, Song KS, Choi GJ. Intraoperative systemic infusion of lidocaine reduces postoperative pain after lumbar surgery: a double-blinded, randomized, placebo-controlled clinical trial. Spine J. 2014 Aug 1;14(8):1559-66. doi: 10.1016/j.spinee.2013.09.031. Epub 2013 Nov 8. PMID 24216403